CLINICAL TRIAL: NCT07034027
Title: Building Emotion Regulation Skills in Young Adults Using an Online Single-Session Intervention: A Randomized Controlled Trial
Brief Title: A Single-Session Intervention Fostering Emotional Nonreactivity
Acronym: Project WAVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00223240
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Emotional Dysregulation

STUDY DESIGN:
Intervention Model Description: This study uses a two-group between-subjects design.
Who Masked: Participant
Masking Description: The measures and intervention will be self-administered, so there is no direct interaction between personnel and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project WAVE (Wise Awareness of Visiting Emotions) (Experimental): The active condition, "Project WAVE," (Wise Awareness of Visiting Emotions) includes 1) an introduction to the program's rationale; 2) psychoeducation about emotion dysregulation, avoidance, and exposure; 3) testimonials from others who describe their experience facing a difficult emotion; 4) an emotion exposure task along with an audio-guided nonreactivity practice; and 5) the creation of a personalized "action plan" usable for continued practice. Project WAVE is designed to take approximately 15-20 minutes.
  Interventions: Behavioral: Project WAVE (Wise Awareness of Visiting Emotions)
- Emotionally Neutral Writing Condition (Placebo Comparator): The control condition is self-administered and structurally similar to Project WAVE (e.g., includes peer narratives and contains a similar number of writing activities). It is designed to control for non-specific aspects of supportive online activities. The activity involves an emotionally neutral writing task (journaling about daily life events). This control condition is designed to take approximately 10-15 minutes.
  Interventions: Behavioral: Emotionally Neutral Writing Control

INTERVENTIONS:
Behavioral: Project WAVE (Wise Awareness of Visiting Emotions) — Project WAVE is an online, self-directed single-session intervention designed to foster emotional nonreactivity skills in young adults aged 18-29.
  Arms: Project WAVE (Wise Awareness of Visiting Emotions)
Behavioral: Emotionally Neutral Writing Control — The control condition is an online, self-directed single-session activity that includes an emotionally neutral writing task.
  Arms: Emotionally Neutral Writing Condition

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a novel online single-session intervention (SSI) designed to improve emotion regulation abilities in young adults (ages 18-29). The active intervention condition, titled "Project WAVE," uses mindfulness skills training and an emotion exposure to teach participants how to cope with distressing emotions. Project WAVE will be evaluated in comparison with another online activity that controls for nonspecific aspects of single-session interventions.

ELIGIBILITY:
* Between the ages of 18 and 29, inclusive
* Self-report comfort in reading and writing in English
* Have access to the Internet through computer, laptop, smartphone, etc.
* Live in the United States or U.S. territories, per IP address
* Provide an endorsement of either "disagree" or "strongly disagree" on at least one of the following three items adapted from the Nonreactivity subscale of the Five Facet Mindfulness Questionnaire: "I was aware of my feelings and emotions without having to react to them"; "I watched my feelings without getting lost in them"; "When I had distressing emotions, I 'stepped back' and was aware of the emotion without getting taken over by it"
* Commit to providing thoughtful answers to the questions asked
* Pass the attention check / bot detection question, "Are you taller than 10 feet?" ("yes," "no," or "unsure") in the initial screener survey

Exclusion Criteria:

* Fail to meet the above-listed inclusion criteria
* Exit the study prior to condition randomization
* Fail to pass data integrity measures

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 545 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Emotion Intolerance Beliefs. | Data will be collected in both conditions at all time points (pre-intervention, immediate post-intervention, and two-week follow-up).
  Emotion intolerance beliefs will be measured using the Emotion Avoidance Questionnaire (EAQ) Beliefs subscale, a five-item self-report measure of a participant's beliefs about their inability to tolerate emotions (Taylor et al., 2004). Participants will rate their agreement with each statement reflecting how they feel "right now" on a five-point scale. A higher score indicates greater levels of negative beliefs about their ability to tolerate emotions.

SECONDARY OUTCOMES:
Perceived Intervention Utility | Data will be collected only in Project WAVE and only at immediate post-intervention.
  Perception of the intervention's utility in teaching nonreactivity will be assessed with the items: "During this activity, to what extent were you able to observe your emotions without getting caught up in them?"; "How much did this activity help you learn how to be nonreactive to distressing emotions?"; "How much do you think being nonreactive to distressing emotions could help you in the future?" (each on a five-point Likert scale ranging from "not at all" to "very much"); and "How likely are you to try being nonreactive to distressing emotions in the future?" (on a five-point Likert scale ranging from "very unlikely" to "very likely"). Participants will also be asked a multi-select question: "Did anything get in the way of being able to complete the nonreactivity practice?" with response options including "It was too hard," "It was confusing," "I didn't find it interesting," "I got distracted," "Something else [write-in]," or "Nothing got in the way."

OTHER OUTCOMES:
Nonreactivity to Emotions | Data will be collected in both conditions at pre-intervention and two-week follow-up.
  Nonreactivity to emotions will be measured using a three-item subset of the Five Facet Mindfulness Questionnaire (FFMQ) Nonreactivity subscale, a seven-item self-report measure of a participant's tendency to react to their emotions (Baer et al., 2008). We are choosing to use a slightly modified three-item subset that has been used in previous research (Galla et al., 2020). For the present purposes, we used "emotions" in place of the original "thoughts or images" because the intervention focuses both on thoughts and body sensations. Participants in both conditions will rate their agreement with each statement reflecting how true each statement was for them over the past two weeks on a five-point scale.
Program Feedback | Data will be collected in both conditions only at immediate post-intervention.
  Similar to previous SSIs (e.g., Schleider et al., 2020), the perceived acceptability of the SSI will be measured using the Program Feedback Scale (PFS). The PFS asks participants to rate agreement with seven statements about the acceptability of the SSI (e.g. "I enjoyed the program") on a five-point scale. A score of 3/5 or above on any given PFS item will be interpreted as an "acceptable" rating on that item (Schleider et al., 2020). Scores are calculated at the item level, and higher scores reflect greater acceptability for each item.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code

REFERENCES:
- [Background] Taylor CT, Laposa JM, Alden LE. Is avoidant personality disorder more than just social avoidance? J Pers Disord. 2004 Dec;18(6):571-94. doi: 10.1521/pedi.18.6.571.54792. PMID 15615668
- [Background] Schleider JL, Dobias M, Sung J, Mumper E, Mullarkey MC. Acceptability and Utility of an Open-Access, Online Single-Session Intervention Platform for Adolescent Mental Health. JMIR Ment Health. 2020 Jun 30;7(6):e20513. doi: 10.2196/20513. PMID 32602846
- [Background] Galla BM, Tsukayama E, Park D, Yu A, Duckworth AL. The mindful adolescent: Developmental changes in nonreactivity to inner experiences and its association with emotional well-being. Dev Psychol. 2020 Feb;56(2):350-363. doi: 10.1037/dev0000877. PMID 31961194
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597